CLINICAL TRIAL: NCT02631655
Title: Study of the Impact of 18F-FDOPA Positon Emission Tomography on Therapeutic Proposals Made at Neurooncology Multidisciplinary Case Conferences
Brief Title: POSitron Emission Imaging Using 18F-FDOPA in Neurooncology
Acronym: POSEIDON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014/60
Record Dates: First submitted 2015-12-05; First posted 2015-12-16 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2020-04

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- device 18FDOPA (Other): impact of device 18F-FDOPA PET on treatment decisions
  Interventions: Other: impact of device 18F-FDOPA PET on treatment decisions

INTERVENTIONS:
Other: impact of device 18F-FDOPA PET on treatment decisions — Imagery device: impact of 18F-FDOPA PET imaging on treatment decisions for patients with high-grade gliomas with an uncertain diagnosis.

SUMMARY:
18F-FDOPA PET is expensive. It is mandatory therefore to assess its impact on the management of patients with high-grade gliomas in order to provide medico-economic justification for its use. The article by the UCLA group showed that 18F-FDOPA modified 41% of management decisions for patients with brain tumors (Walter JNM 2012). However, this study comprised 58 patients, combined primary and recurring tumors, and was based on questionnaires sent out to referring physicians. A targeted study is needed, therefore, to make a prospective multicenter assessment of the contribution of this technique in the context of high-grade glial tumors and neurooncology MCCs.

DETAILED DESCRIPTION:
Current treatment of high-grade glioma combining surgery, radiotherapy and chemotherapy has enhanced overall survival during the past 10 years, notably thanks to the " Stupp " protocol using Temozolomide. At tumor evaluation and post-treatment follow-up, decisions regarding management (change, discontinuation or continuation of treatment) are discussed during multidisciplinary case conferences (MCC) between neurooncology specialists and are generally based primarily on MRI data. New treatment strategies are more effective on tumor tissue but also affect the adjacent healthy tissue. These phenomena give rise to complex MRI changes which can make it more difficult to perform differential diagnoses between tumor recurrence and treatment sequellae, such as radionecrosis and pseudoprogression. Alternatively, they can conceal effective tumor progression (appearance of pseudoresponse under antiangiogenics). Classical MRI interpretation criteria have evolved to take these phenomena into account (RANO criteria) and are now supplemented by new MRI data (perfusion and diffusion imaging, spectroscopy). Nonetheless, cases involving an uncertain recurrence diagnosis are still frequent. PET imaging has also shown very good results in differential diagnosis between posttreatment changes. Fluorodeoxyglucose-18-F (18FDG) can be used for glioma follow-up (Varrone EJNMMI 2009) but produces false positives during follow-up. In this setting, over-expression of amino acid transporter LAT-1 in brain tumors makes amino acids or marked analogs more suitable for PET imaging of glial tumors. C-11 methionine and 18F-FET can be used, but 18F-FDOPA is currently the only radiopharmaceutical agent to have received marketing authorization in France. Recently, the UCLA group demonstrated that 18F-FDOPA could modify the intended management of 41% of patients with brain tumors . The present projects aims to assess the impact of 18F-FDOPA PET imaging on decisions taken by neurooncology MCCs for the management of patients already treated for high-grade gliomas.

Expected benefits for patients and in terms of Public Health High-grade gliomas are the commonest and most aggressive brain tumors. Current therapy combining several treatments (surgery, radiotherapy, radiosurgery and chemotherapy) has improved overall patient survival during the past 10 years. Nevertheless, tumor recurrence accounts for a median survival of approximately only 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with high-grade glioma
* Patient whose file has been submitted to the neurooncology MCC for follow-up after initial treatment and for whom there is a diagnostic doubt
* Age > 18 years
* Patient has been informed and has signed informed consent for the study

Exclusion Criteria:

* Patient presenting comorbidities or allergies on account of which MRI or 18F-FDOPA PET would be contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-12; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
percentage of modified therapeutic decisions connected to the data supplied by 18F-FDOPA PET | up to 3 years

SECONDARY OUTCOMES:
Percentage of variation in the confidence level of diagnosis incorporating 18F-FDOPA PET findings (reduced, unchanged, increased). | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jacques DARCOURT, PHD, Study Director — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France